CLINICAL TRIAL: NCT03776409
Title: Comparison of the Nephrotoxicity of Vancomycin in Combination With Piperacillin/Tazobactam or Other Beta-lactams in Critically Ill Patients: A Retrospective, Multicenter Study in China
Brief Title: Safety and Efficacy of Vancomycin Plus Beta-lactams
Acronym: SEVPB
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2018LSK-169
Record Dates: First submitted 2018-12-06; First posted 2018-12-14 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2018-12

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Vancomycin; Piperacillin; Tazobactam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vancomycin plus piperacillin/tazobactam: Critically ill patients who received the combination of VAN (vancomycin) and PTZ (piperacillin/tazobactam) for at least 48 hours during an ICU (intensive care unit) admission, had a baseline serum creatinine (Scr) concentration value within 24 hours of hospital admission.The dosage and frequency of VAN and PTZ were adjusted based on clinical practice and patient characteristics. This is an observational study without any intervention.
  Interventions: Drug: vancomycin plus piperacillin/tazobactam
- vancomycin plus other beta-lactams: Critically ill patients who received the combination of VAN (vancomycin) and other beta-lactams (cefoperazone/sulbactam, meropenem, imipenem/siastatin, ceftriaxone, ceftazidime, et al) for at least 48 hours during an ICU (intensive care unit) admission, had a baseline serum creatinine (Scr) concentration value within 24 hours of hospital admission.The dosage and frequency of VAN and other beta-lactams were adjusted based on clinical practice and patient characteristics. This is an observational study without any intervention.
  Interventions: Drug: vancomycin plus other beta-lactams

INTERVENTIONS:
Drug: vancomycin plus piperacillin/tazobactam — Patients in intensive care unit who received the combination of VAN(vancomycin) and PTZ (piperacillin/tazobactam) for at least 48 hours, had a serum creatinine level measured in the 24-hour of hospital admission.The dosage and frequency of VAN and PTZ was adjusted based on clinical practice and patient characteristics.
  Groups: vancomycin plus piperacillin/tazobactam
Drug: vancomycin plus other beta-lactams — Patients in intensive care unit who received the combination of VAN (vancomycin) and other beta-lactams (cefoperazone/sulbactam, meropenem, imipenem/siastatin, ceftriaxone, ceftazidime, et al) for at least 48 hours, had a baseline serum creatinine (Scr) concentration value within 24 hours of hospital admission.The dosage and frequency of VAN and other beta-lactams were adjusted based on clinical practice and patient characteristics.
  Groups: vancomycin plus other beta-lactams

SUMMARY:
The combination of vancomycin and piperacillin-tazobactam has been associated with an increased risk of acute kidney injury (AKI) in non-critically ill patient populations, but it is still unknown if this association exists in critically ill patients. The objective of this study is to compare AKI and efficacy of vancomycin plus piperacillin-tazobactam or beta-lactams.

DETAILED DESCRIPTION:
The combination of vancomycin and piperacillin-tazobactam has been associated with an increased risk of acute kidney injury (AKI) in non-critically ill patient populations, but limited data regarding this association exists in critically ill patients. The objective of this study is to compare AKI and efficacy of vancomycin plus piperacillin-tazobactam or beta-lactams.

This is a multicenter, retrospective cohort study. Patients from the retrospective cohort will be divided into 2 groups based on the combination regimen received . Patients who meet the inclusion and exclusion criteria will be included in our registry. As a non-intervention study, these information as below will be collected: basic demographics, diagnosis, concomitant nephrotoxic and other antibiotic medications, serum creatine levels, vancomycin concentrations, and indication for antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* admitted to intensive care unit
* received the combination of vancomycin and beta-lactams for at least 48 hours
* had a serum creatinine level measured within 24-hour hospital admission
* had at least one VAN level drawn while receiving a combination of study antibiotics

Exclusion Criteria:

* pregnancy or lactating patients
* admission to the intensive care unit during administration or within 72 hours of completing the antibiotics
* had end-stage renal disease
* died within 48 hours of combination antibiotic therapy initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
AKI(acute kidney injury) | from 24 hours after the start of the combination until discharge up to one month
  the incidence of acute kidney injury
clinical efficacy | from 24 hours after the start of the combination until discharge up to one month
  microbial eradication

SECONDARY OUTCOMES:
the length of hospital stay | from hospital admission to discharge up to one month
duration of AKI | the time from AKI onset to resolution of AKI up to one month
onset of AKI | the first occurence of AKI after starting concomitant antimicrobial use up to one month
whether renal function return to baseline or not | from AKI onset to resolution of defined AKI up to one month
  whether defined AKI was resoluted or not
major acute kidney events at 30 days (MAKE30) | MAKE30 is assessed 30 days following AKI diagnosis
  MAKE30 is assessed 30 days following AKI diagnosis, which is a composite outcome of death, new dialysis, and worsened renal function.
vancomycin trough value assessment | from hospital admission to discharge up to one month
  assess the impact of vancomycin exposures on development of AKI

CONTACTS AND LOCATIONS:
Overall Officials: Yalin Dong, Ph.D, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No